CLINICAL TRIAL: NCT03731130
Title: Radiation or Chemoradiation Followed by Surgery in Patients With Rectal Cancer
Brief Title: Prospective Observational Trial to Evaluate Quality of Life After Neoadjuvant Radiation or Chemoradiation Followed by Surgery in Patients With Rectal Cancer
Acronym: NEOCARE
Status: Recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Falk Roeder, Consultant, Ludwig-Maximilians - University of Munich
Other Study IDs: V1 10.07.2018
Record Dates: First submitted 2018-10-17; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Rectal Cancer; Quality of Life; Radiation Therapy; Chemoradiation
Keywords: rectal cancer; quality of life; neoadjuvant; radiation therapy; chemoradiation
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neoadjuvant short term radiation: Treatment with neoadjuvant short term radiation therapy (5x5 Gy) followed by surgery. Quality of life will be assessed using the EORTC QLQ C30 and EORTC QLQ CR 29 questionaire.
  Interventions: Other: EORTC QLQ C30; Other: EORTC QLQ CR29
- neoadjuvant long-term chemoradiation: Treatment with neoadjuvant Long-term chemoradiation followed by surgery. Quality of life will be assessed using the EORTC QLQ C30 and EORTC QLQ CR 29 questionaire
  Interventions: Other: EORTC QLQ C30; Other: EORTC QLQ CR29

INTERVENTIONS:
Other: EORTC QLQ C30 — standardized questionaire
Other: EORTC QLQ CR29 — standardized questionaire

SUMMARY:
Observational study to evaluate longitudinal quality of life according to standardized EORTC questionaires as well as functional Outcome, oncological outcome and toxicity in patients treated with neoadjuvant short term radiation or long-term chemoradiation followed by surgery

DETAILED DESCRIPTION:
Observational study to evaluate longitudinal quality of life in patients treated with neoadjuvant short-course Irradiation or neoadjuvant Long-Course chemoradiation followed by surgery. QoL will be evaluated by standardized EORTC questionaires QLQ C30 and CR29. Acute and late toxicity will be assessed according to CTCAE 4.03. Oncological Outcome will be assessed with regard to local and distant Control, Patterns of recurrence, freedom from Treatment failure and Overall survival. Correlations of physicians- and Patient-assessed functional outcomes are planned.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven rectal Cancer without distant metastases
* indication for neoadjuvant Radiation or chemoradiation therapy according to multidiciplinary Evaluation
* age >=18 years
* written informed consent
* ability to answer the standardized questionaires according to the treating physician

Exclusion Criteria:

* age < 18 years
* prior systemic therapy with regard to rectal Cancer
* distant metastasis
* second malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: see eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-10-05 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
QoL (EORTC QLQC30) absolute values and change over time | short-term radiation: day 0, end of week 1, 14, 27, 53, 105, 157, 209, 261, long-term chemoradiation: day 0, end of week 6, 14, 27, 40, 66, 118, 170, 222, 274
  Quality of life measured by EORTC questionaires QLQC30 in absolute values at different time points and change over time
QoL (EORTC QLQCR29) absolute values and change over time | short-term radiation: day 0, end of week 1, week 14, 27, 53, 105, 157, 209, 261, long-term chemoradiation: day 0, end of week 6, 14, 27, 40, 66, 118, 170, 222, 274
  Quality of life measured by EORTC questionaires QLQCR29 in absolute values at different time points and change over time

SECONDARY OUTCOMES:
acute toxicity | short-term radiation: day 0, end of week 1, long-term chemoradiation: day 0, end of week 6, 14
  acute toxicity by Radiation or chemoradiation according to CTCAE 4.03
late toxicity | short-term radiation: end of week 27, 53, 105, 157, 209, 261, long-term chemoradiation: end of week 27, 40, 66, 118, 170, 222, 274
  late toxicity according to CTCAE 4.03
local control | short-term radiation: day 0, end of week 1, 14, 27, 53, 105, 157, 209, 261, long-term chemoradiation: day 0, end of week 6, 14, 27, 40, 66, 118, 170, 222, 274
  Absence of local regrowth
distant control | short-term radiation: day 0, end of week 1, 14, 27, 53, 105, 157, 209, 261, long-term chemoradiation: day 0, end of week 6, 14, 27, 40, 66, 118, 170, 222, 274
  Absence of distant metastases
freedom from Treatment failure | short-term radiation: day 0, end of week 1, 14, 27, 53, 105, 157, 209, 261, long-term chemoradiation: day 0, end of week 6, 14, 27, 40, 66, 118, 170, 222, 274
  Absence of local or distant relapse
Overall survival | short-term radiation: day 0, end of week 1, 14, 27, 53, 105, 157, 209, 261, long-term chemoradiation: day 0, end of week 6, 14, 27, 40, 66, 118, 170, 222, 274
  Absence of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Falk Roeder, MD, Principal Investigator — Ludwig-Maximilians Universität München
Locations (1):
- Department of Radiation Oncology, University Hospital, LMU Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No